CLINICAL TRIAL: NCT00841165
Title: Randomized Trial of Carbon Monoxide Elimination Kinetics With Oxygen Delivered by Continuous Positive Airway Pressure Compared to Face Mask
Brief Title: Carbon Monoxide Monitoring and Emergency Treatment
Acronym: COMET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Vermont (Other)
Responsible Party: Dr. Kalev Freeman, Faculty Sponsor, Department of Surgery, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHRMS 09-056
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-04

CONDITIONS: Carbon Monoxide Poisoning
Keywords: Carbon Monoxide Toxicity; Carbon; Monoxide; Poisoning; Toxicity; Treatment; CPAP; Hyperbaric; Oxygen
MeSH Terms: conditions — Carbon Monoxide Poisoning; Poisoning | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants in this arm are treated with Continuous Positive Airway Pressure at 5cm H2O and 100% oxygen
  Interventions: Device: Continuous Positive Airway Pressure
- 2 (Active Comparator): Participants in this arm receive standard of care therapy- oxygen via a non-rebreather mask
  Interventions: Device: Non-rebreather oxygen mask

INTERVENTIONS:
Device: Continuous Positive Airway Pressure — Full face CPAP at 5cm H2O and 100% oxygen
  Arms: 1
Device: Non-rebreather oxygen mask — Oxygen administered through a non-rebreather mask
  Arms: 2

SUMMARY:
Carbon monoxide (CO) has been called a "silent killer", and those patients who survive CO poisoning are at risk of neurological damage, which may be permanent. CO is a leading cause of unintentional poisoning deaths in the United States, and the odorless gas results in an estimated average of 20,636 emergency department (ED) visits each year. Oxygen is the antidote for CO poisoning, and it acts both by attenuating toxic effects and enhancing elimination. A fractional inspired concentration of oxygen (FiO2) of 0.7 to 0.9 may be achieved by administration of 100% oxygen delivered using a reservoir with a facemask that prevents rebreathing. Hyperbaric oxygen therapy may provide added benefit for patients with CO poisoning, but this therapy is unavailable in many parts of the United States including Vermont. Use of a continuous positive airway pressure (CPAP) mask may achieve an FiO2 of 1.0, but the effects of delivering an FiO2 of 1.0 compared to 0.7 in CO poisoning are unknown. CPAP, by comparison, is inexpensive, portable, and available in most EDs. In this study, the investigators are testing the hypothesis that oxygen delivered by CPAP will improve both CO washout kinetics and functional outcomes, compared to the standard therapy of oxygen delivered by non-rebreathing facemask. Specific Aim 1 will provide toxicokinetic data to support a potential benefit in the use of CPAP for CO poisoning, by comparing CO elimination kinetics in response to oxygen therapy delivered by non-rebreathing facemask versus CPAP. The 20 patients expected in our first year will provide adequate power to detect a 20% fall in half-time of CO elimination. While CPAP may increase CO washout rates, as predicted in Specific Aim 1, demonstration of real functional benefit will be tested in Specific Aim 2. This Aim seeks to determine functional (neuropsychological) outcomes in patients with CO poisoning treated with oxygen therapy delivered by non-rebreathing facemask versus CPAP. Data showing a therapeutic benefit from CPAP in CO poisoning would have clinical implications. Compared to hyperbaric oxygen therapy, CPAP therapy can begin earlier, including the pre-hospital setting, for patients with known exposure. With the frequent nature of CO poisoning and the widespread availability of CPAP, a potential benefit could lead to improved outcomes for the 20,000+ patients who present to EDs annually.

ELIGIBILITY:
Inclusion Criteria:

* Elevated Carboxyhemoglobin Level (non-smokers >8%, smokers >12%)
* 18 years of age or older
* Able to provide informed consent as assessed by Attending Emergency Physician

Exclusion Criteria:

* Requires daily medication for active lung disease
* Altered mental status
* Hemodynamically unstable
* Requires transfer to ICU or hyperbaric oxygen facility
* Previous enrollment in the study
* No concurrent acute psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Half life of Carboxyhemoglobin | Every 15 minutes during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kalev Freeman, MD, PhD, Study Director — University of Vermont
Locations (1):
- Fletcher Allen Health Care, Burlington, Vermont, United States

REFERENCES:
- [Background] Bruce MC, Bruce EN. Analysis of factors that influence rates of carbon monoxide uptake, distribution, and washout from blood and extravascular tissues using a multicompartment model. J Appl Physiol (1985). 2006 Apr;100(4):1171-80. doi: 10.1152/japplphysiol.00512.2005. Epub 2005 Dec 8. PMID 16339350
- [Background] Bruce EN, Bruce MC. A multicompartment model of carboxyhemoglobin and carboxymyoglobin responses to inhalation of carbon monoxide. J Appl Physiol (1985). 2003 Sep;95(3):1235-47. doi: 10.1152/japplphysiol.00217.2003. Epub 2003 May 16. PMID 12754170
- [Background] Weaver LK. Clinical practice. Carbon monoxide poisoning. N Engl J Med. 2009 Mar 19;360(12):1217-25. doi: 10.1056/NEJMcp0808891. No abstract available. PMID 19297574